CLINICAL TRIAL: NCT05842746
Title: Efficacy and Safety of Elemene Plus Stupp Protocol Versus Stupp Protocol Alone for Newly-diagnosed Glioblastoma: A Multi-center Phase II Randomized Controlled Trial
Brief Title: Elemene Plus Stupp Protocol Versus Stupp Protocol Alone for Newly-diagnosed Glioblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K3649-I-23PJ571
Record Dates: First submitted 2023-04-09; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma, IDH-wildtype
MeSH Terms: conditions — Glioblastoma | interventions — elemene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stupp Protocol (Placebo Comparator): Patients receive maximal safe tumor resection, concurrent radiochemotherapy with TMZ, and adjuvant TMZ (the Stupp Protocol). Placebo that has the same appearance and flavor with Elemene is given 20ml orally, three times a day for 28 consecutive days (as one cycle) for 6 cycles, during the phase of adjuvant TMZ administration.
  Interventions: Drug: Placebo
- Ele-Stupp Protocol (Experimental): Patients receive maximal safe tumor resection, concurrent radiochemotherapy with TMZ, and adjuvant TMZ (the Stupp Protocol). Elemene is given 20ml:176mg orally, three times a day for 28 consecutive days (as one cycle) for 6 cycles, during the phase of adjuvant TMZ administration.
  Interventions: Drug: Elemene

INTERVENTIONS:
Drug: Elemene — Elemene of 20ml is given orally, three times a day, for 28 consecutive days (as a cycle), for 6 cycles.
  Arms: Ele-Stupp Protocol
Drug: Placebo — Placebo (with the same appearance and flavor with Elemene) of 20ml is given orally, three times a day, for 28 consecutive days (as a cycle), for 6 cycles.
  Arms: Stupp Protocol

SUMMARY:
The goal of this phase II randomized clinical trial is to compare the safety and efficacy of Elemene plus Stupp Protocol (the new protocol) and Stupp Protocol alone (the standard protocol) in patients with newly-diagnosed glioblastomas (ndGBMs). The main questions to answer are:

* Whether the new treatment protocol (Elemene plus Stupp Protocol) is clinically safe for ndGBM patients.
* Whether the new treatment protocol (Elemene plus Stupp Protocol) brings better survival benefits for ndGBM patients compared to the standard-of-care Stupp Protocol.

Study participants will be enrolled in 5 hospitals in China and randomly assigned to receive either the new protocol or the standard protocol. The overall survival (OS) rate in the 12th month, the progression-free survival (PFS) rate in the 6th month, OS, PFS, and adverse events assessed by the CTCAE (Common Terminology Criteria for Adverse Events) will be evaluated for all patients.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is a WHO grade 4 adult-type diffuse glioma and the most common malignant, primary brain tumor with a 5-year overall survival (OS) of only ~5% in real-world studies. The Stupp Protocol, consisting of fractionated focal irradiation in daily fractions of 2 Gy given 5 days/week for 6 weeks (a total of 60 Gy), plus concomitant daily temozolomide (TMZ, 75 mg/m2/day, 7 days/week from the first to the last day of radiotherapy) after maximal safe tumor resection, followed by six cycles of adjuvant TMZ (150-200 mg/m2/day for 5 days during each 28-day cycle), has been adopted as the standard of care for patients with newly-diagnosed GBMs (ndGBMs) since 2005.

However, there have been no other treatment modalities except for tumor treating fields (TTFields) that have brought survival benefits for ndGBM patients during the past two decades. Since TTFields therapy is super expensive (about 1 million yuan/0.15 million dollars per year) and fewer than 10% of ndGBM patients can afford it around the globe, the Stupp Protocol is still being used as the first-line and the most widely-adopted treatment option for ndGBM patients around the world.

Elemene, a Chinese anti-tumor medicine extracted from the plant Curcuma Wenyujin, has been isolated as a monomeric drug and has a broad-spectrum anti-tumor effect in various cancers, such as lung cancer, breast carcinoma, leukemia, and ovarian cancer. In recent years, its application in GBMs as revealed in the preliminary retrospective studies published in Chinese Journals and a few English Journals have shown survival benefits with acceptable toxicity. Elemene can pass through the blood-brain barrier because of its small molecular weight and lipid solubility and has synergistic anti-tumor effects with TMZ and radiotherapy for GBM patients. Several in vitro studies also have shown that Elemene could inhibit GBM cell proliferation, promote cell differentiation, and induce cancer cell apoptosis.

All these findings from the above studies have indicated the potential survival benefits of Elemene in treating ndGBMs. However, so far, no clinical trials have tested the efficacy and safety of the new treatment protocol (Elemene added to the Stupp Protocol) for ndGBMs compared with the conventional Stupp protocol.

In this study, the investigators aimed to launch a multi-center, phase II, randomized, controlled clinical trial to test the safety and efficacy of Elemene plus Stupp Protocol compared with Stupp Protocol alone for ndGBM patients.

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed supratentorial glioblastoma, IDH-wildtype, WHO grade 4
* male or female adult patients < 70 years old
* Karnofsky performance status (KPS) score higher or equal to 60
* a minimum life expectancy of 12 weeks
* adequate bone marrow function (white blood cell ≥ 2.0 × 10^9/L, neutrophils ≥ 1.5 × 10^9/L, hemoglobin ≥ 90 g/L, and platelets ≥ 100 × 10^9/L)
* adequate hepatic function (direct bilirubin and indirect bilirubin ≤ 1.5 mg/dL, and alanine aminotransferase [ALT] and aspartate aminotransferase [AST] < 4 times the upper limit of normal)
* adequate renal function (creatinine < 80 umol/L)
* adequate coagulation function (international normalized ratio [INR] ≤ 1.3)
* voluntary to participate in this trial, complete all pre-specified treatment regimens, and complete required follow-up

Exclusion Criteria:

* unwilling to participate or accept the pre-specified treatment regimen and required follow-up schedule
* prior treatment (surgery, radiotherapy, chemotherapy) for glioblastoma
* pregnant or lactating patients
* allergic to Elemene and its components
* severe liver and kidney dysfunction, coagulation disorders, or decreased hematopoietic ability
* serious infection
* serious hyperlipidaemia
* medical illness or psychosocial circumstance that may compromise participant safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The overall survival (OS) rate in the 12th month (12m-OS) | 12th month after randomization
  The rate of patients who are still alive in the 12th month after randomization

SECONDARY OUTCOMES:
The overall survival (OS) | From randomization to death, assessed up to 24 months
  The survival time from randomization to death from any cause
The progression-free survival (PFS) | From randomization to objective tumor progression or death, assessed up to 24 months
  The survival time from randomization to objective tumor progression or death
The progression-free survival (PFS) rate in the 6th month (6m-OS) | 6th month after randomization
  The rate of patients who have no objective tumor progression in the 6th month after randomization
Adverse events | From randomization to death, assessed up to 24 months
  Adverse events evaluated using the CTCAE version 4.03

OTHER OUTCOMES:
Subgroup analyses for primary and secondary outcomes | From randomization to death, assessed up to 24 months
  Subgroups to be divided by sex, age, molecular alterations, KPS score, and extent of resection.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Ma, MD, Study Chair — Peking Union Medical College Hospital; Yu Wang, MD, PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) can be made available upon publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication.
Access Criteria: Via communication with the corresponding authors.